CLINICAL TRIAL: NCT06629545
Title: Comparison of Passive Ultrasonic and Sonically Activated Irrigation Methods in the Treatment of Apical Periodontitis: Evaluation of PGE2, NO and IL-6 Levels
Brief Title: The Efficacy of Two Different Irrigation Methods on PGE2, NO and IL-6 Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Seyda Ersahan, DDS, PhD, Seyda Ersahan, Clinical Associate Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023
Record Dates: First submitted 2024-10-01; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-06

CONDITIONS: Apical Periodontitis; Inflammatory Markers
Keywords: apical periodontitis; passive ultrasonic irrigation; Sonically Activated Irrigation; Gingival crevicular fluid; PGE; IL-6
MeSH Terms: conditions — Periapical Periodontitis | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Passive ultrasonic irrigation (Experimental): The irrigation solution was agitated by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device.
  Interventions: Other: irrigation activation with PUI
- Sonic activated irrigation (Experimental): The irrigation solution was agitated by a suitable-size activator tip (#25/.04) attached to an EndoActivator sonic handpiece (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA).
  Interventions: Other: irrigation with sonic activation
- Control group (No Intervention): Pre-treatment GCF (preGCF) samples were collected for all participants

INTERVENTIONS:
Other: irrigation activation with PUI — The irrigation solution was used by adapting an ultrasonic tip (IRRI S 21/25; VDW, Munich, Germany) to an ultrasonic device. The power setting of the ultrasonic device was 30% (VDW Ultra; VDW, Munich, Germany). The tip was activated a total of three times, with each cycle lasting 20 s and involving the use of 1 ml of 2.5% NaOCl. Then, 2 ml of 17% EDTA solution was activated for 1 min as describe above. The ultrasonic tip was placed 1 mm behind the working length without touching the canal walls.
  Arms: Passive ultrasonic irrigation
Other: irrigation with sonic activation — A suitable-size activator tip (#25/.04) attached to an EndoActivator sonic handpiece (Dentsply Tulsa Dental Specialties, Tulsa, OK, USA) was inserted into the canal 1 mm short of the working length. 3 ml of 2.5% NaOCl solution was activated in three periods of 20 s (1 ml of 2.5% NaOCl in each cycle). Then, the same procedure was repeated with 2 ml of 17% EDTA solution.
  Arms: Sonic activated irrigation

SUMMARY:
Today, debates about the effectiveness of Passive Ultrasonic Irrigation (PUI) and Sonically Activated Irrigation (SAI) techniques used to increase the success of endodontic treatment in chronic apical periodontitis (AP) are still ongoing.

In this study, the effectiveness of PUI and SAI systems was investigated in AP patients with similar infection burden and periapical lesion size (PLS) based on changes in prostaglandin E2 (PGE2), nitric oxide (NO) and interleukin-6 (IL-6) levels, which are important biomarkers of inflammatory response in gingival crevicular fluid (GCF) samples.

The study was planned as a single-center cross-sectional analytical study. A total of 60 patients with AP requiring root canal treatment [PUI (n:30) and SAI (n:30)] and 30 healthy controls were included in the study between January and June 2024. Demographic characteristics of the patients as well as clinical and radiographic findings (PLS and PAI score) were recorded. GCF (preGCF), PGE2, NO and IL-6 levels were measured in all participants before irrigation. The same procedure was repeated in GCF samples 1 week after treatment (postGCF), except for the control group. In addition, 1st order most commonly seen bacteria (FMCB) typing was performed on swab samples taken from the root canals of the patients.

DETAILED DESCRIPTION:
The diagnosis was established according to the patient's history, clinical inspection including palpation, tenderness to percussion, pulpal sensitivity testing, and radiographic examination. Demographic characteristics of the participants (age, gender, chronic disease status, etc.) as well as clinical and radiographic findings [pain level, number of crowns (NC), number of fillings (NF), number of root canal fillings (NRC), and number of missing teeth (NMT)] were recorded. Panoramic and periapical dental radiographs were taken. The presence of radiolucent images associated with the periapical region and radiographic bone loss were evaluated. Radiographs were examined with the help of Kodak Dental Imaging Software. The presence of periapical radiolucency without periodontal disease was considered sufficient criteria for the diagnosis of AP. The largest diameter of the lesion was measured on preoperative periapical radiographs and recorded as periapical lesion size (PLS). In addition, periapical index (PAI) score defined by Ørstavik et al (Ørstavik et al., 1986) and abscess scoring based on the periapical index (AS-PAI) were recorded for patients with AP. AS-PAI was determined as follows: AS-PAI-0 if PAI<5, AS-PAI-1 if only 1 tooth with PAI 5 and AS-PAI-2 if >2 teeth with PAI 5

ELIGIBILITY:
Inclusion Criteria:

For control group

* People who come for a check-up, are healthy in terms of dental and periodontal health, do not have any systemic acute or chronic disease (such as infection, kidney disease, cardiovascular disease, inflammatory and rheumatic disease, diabetes and local or widespread tissue damage) and have similar values in terms of gender, age and weight to the study groups, For experimental groups
* Being systemically healthy,
* Patients between the ages of 18-65,
* Those having a PAI score of 3-5 For both study and control groups
* The volunteer wishes to participate in the research by signing the 'Informed Consent Form'.

Exclusion Criteria:

* Those who have used nonsteroidal anti-inflammatory drugs and/or immunosuppressive drugs, steroids in the last 48 hours as this may affect the test results, and those who have a history of using high doses of biotin vitamin as this may affect the test results,
* Those who were either pregnant, lactating, morbidly obese, presence of malignancy, presence of concomitant infection other than AP, presence of acute or chronic inflammatory disease,
* Those with periodontal disease (with periodontal pockets and attachment levels exceeding 4 mm.),
* Those having inadequate crown structures for isolation with a rubber dam,
* Those with a history of previous endodontic treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
ELISA Analysis of Biochemical Parameters | Up to 36 weeks
  ELISA assay was performed to measure preGCF and postGCF-PGE2, NO and IL-6 levels

SECONDARY OUTCOMES:
Genomic DNA isolation and measurement of DNA concentration | Up to 36 weeks
  Pretreatment bacteria number and bacteria species of samples taken from root canals measured via PCR and Sanger sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Ersahan, Assoc.Prof., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: starting 6 months after publication
Access Criteria: The investigators want to share IPD including all ddPCR and ELISA results with all researchers